CLINICAL TRIAL: NCT06371300
Title: Photobiomodulation of the Ocular Surface and Eyelids With Different Wavelengths: REd vs BluE Light (REBEL)
Brief Title: Photobiomodulation With REd vs BluE Light (REBEL)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HLS21156
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye Syndromes; Meibomian Gland Dysfunction; Blepharitis
Keywords: Low-level light therapy
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction; Blepharitis

STUDY DESIGN:
Intervention Model Description: Each participant is randomised to either of 3 groups: Red light only group, red plus blue light group, or sham treatment group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Red light only group (Active Comparator): LLLT will be administered using the Espansione Group Ltd Eye-light unit. LLLT consisting of a wearable facial mask with red light emitting diodes (LEDs) is administered for 30 minutes.
  Interventions: Device: Red LLLT
- Red plus blue light group (Experimental): LLLT consisting of a wearable facial mask with red LEDs is administered for 15 minutes, followed by a mask with blue LEDs for another 15 minutes.
  Interventions: Device: Red LLLT; Device: Blue LLLT
- Sham treatment group (Sham Comparator): Sham treatment will be administered by using facial mask with red LEDs emitting at less than 10% fluence power output for 15 minutes, followed by a mask with blue LEDs emitting at less than 10% fluence power output for another 15 minutes.
  Interventions: Device: Sham Red LLLT; Device: Sham Blue LLLT

INTERVENTIONS:
Device: Red LLLT — Mask with LEDs emitting at wavelengths of 633nm to facial and eyelids region with their eyes closed
  Arms: Red light only group; Red plus blue light group
Device: Blue LLLT — Mask with LEDs emitting at wavelengths of 428nm to facial and eyelid regions with their eyes closed
  Arms: Red plus blue light group
Device: Sham Red LLLT — Mask with LEDs emitting at wavelengths of 633nm, but with <10% fluence power output, to facial and eyelids region with their eyes closed
  Arms: Sham treatment group
Device: Sham Blue LLLT — Mask with LEDs emitting at wavelengths of 428nm, but with <10% fluence power output, to facial and eyelids region with their eyes closed
  Arms: Sham treatment group

SUMMARY:
The use of photobiomodulation or low-level light therapy (LLLT) in the ophthalmic field stemmed from dermatology which has shown impact on skin blood flow and regeneration. There has been a rise in clinical interest with emerging evidence in the benefits of photobiomodulation in managing chronic inflammatory conditions such as dry eye disease including improvements in ocular discomfort symptoms, tear film stability and tear volume. Despite the observed clinical benefits, limited research has been done to compare photobiomodulation utilising different wavelengths, as most research on dry eye disease has focused on red wavelengths. It has been purported that blue wavelengths may disrupt microbial growth while red wavelengths stimulate energy production and hence increase heat in the affected tissues, although research into these differential impacts at the ocular surface and external eye has been limited. Hence, the aim of this exploratory clinical trial is to compare the impact of using LLLT incorporating red versus blue wavelengths on eyelid haemodynamics and microbiome, as well as conventional ocular surface measures of patients with dry eye disease and blepharitis (inflammation of the eyelids).

Participants with dry eye disease, oil gland disruption and blepharitis will receive 3 treatments with these LLLT, each separted by 1 week apart, and followed up to 1 month after the final treatment session. Participants will be randomised to either of 3 groups: Red light only group, Red + Blue light group, or a sham treatment group.

DETAILED DESCRIPTION:
This study will be a randomized, double-masked, exploratory clinical study to assess the potential difference in impact between the two wavelengths used for LLLT. The whole study involves a total of 4 visits (consisting of 3 treatment visits, and 1 follow-up visit). All visits will be conducted at the Aston Dry Eye Clinic in Aston University, Birmingham, United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with dry eye disease symptoms (Ocular Surface Disease Index questionnaire (OSDI) score ≥ 13 or Dry Eye Questionnaire (DEQ5) score > 6) and signs (tear film instability measured with non-invasive tear break-up time < 10 s or ocular surface damage measured using special dyes placed on the front surface of the eyes that temporarily stains any aggravated or damaged cells: > 5 corneal spots, > 9 conjunctival spots or lid margin staining ≥ 2mm in length and ≥ 25% in width)
* Individuals need to also have Meibomian gland dysfunction. The diagnosis of Meibomian gland dysfunction depends on how many of 5 glands in the central lower eyelid can express oil, and the quality of the oil. A diagnosis is made if there is decreased expressibility (grade 1-3 on the Pflugfelder scale) and reduced quality of oil (grade 1-3 on Bron scale). Any presence of gland blockage and/or loss of oil glands grade 1 to grade 4 of either eyelid [Pult and Reide-Pult, 2013]) will also justify a diagnosis of Meibomian gland dysfunction.
* Individuals will also need to have ocular demodicosis, diagnosed by clinical observation on slit lamp biomicroscope based on signs including collarettes around the base of lashes, visible Demodex tails, or excessive pouting of lash follicles in those with good lid hygiene where Demodex was confirmed by secondary means such as visible Demodex tails.
* Age ≥ 18 years, male or female
* Able to provide written consent in English
* Able to attend a total of 4 visits: 3 treatment visits and followed up for 1 month after final treatment

Exclusion Criteria:

* Pregnancy
* Ocular light-based therapies including intense pulsed light (IPL) or LLLT treatment within the past 1 month or during study period in addition to those provided in the study
* Contact lens wear in the past 2 weeks or during study period
* Other active ocular surface diseases or history of ocular surgery or corneal infections the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Bacterial Colony to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Measure of number of bacterial colonisation obtained from eyelid swabs

SECONDARY OUTCOMES:
Change from Baseline in Visual Acuity to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Subjective measure of visual acuity using Logarithm of the Minimum Angle Resolution (logMAR) scoring, ranging from -0.30 which signify the ability to be able to resolve the smallest letters, to 1.00 which signify the ability to resolve only the largest letters
Change from Baseline in Non-invasive Tear Break Up Time to the Final Follow-up 1 Month After Final Treatment Session | Baseline and 1 month after final treatment session
  Measure of the stability of tears and how fast the tears evaporate in seconds using the Oculus Keratograph 5M instrument. An average of 3 measurements is obtained.
Change from Baseline in Blink Rate to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Manual subjective count of the number of blinks using the Oculus Keratograph 5M instrument.
Change from Baseline in Tear Meniscus Height to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Measure of the volume of tears in mm using the Oculus Keratograph 5M instrument. An average of 3 measurements is obtained.
Change from Baseline in Lipid Layer Pattern Grading to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Subjective grading of the appearance of the lipid layer pattern as a surrogate measure of its thickness using the Oculus Keratograph 5M instrument. This ranges from Grade 1 indicating very thin lipid layer to Grade 6 indicating very thick lipid layer.
Change from Baseline in Bulbar Conjunctival Hyperaemia to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Automated objective grading of the bulbar conjunctival redness using the Oculus Keratograph 5M instrument. This ranges from Grade 0 indicating no redness to Grade 4 indicating substantial redness.
Change from Baseline in Limbal Conjunctival Hyperaemia to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Automated objective grading of the limbal conjunctival redness using the Oculus Keratograph 5M instrument. This ranges from Grade 0 indicating no redness to Grade 4 indicating substantial redness.
Change from Baseline in Blood Flow to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Measure of blood flow using laser doppler flowmetry instrument.
Change from Baseline in Saponification Grading to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Measure of saponification on a scale of 0 (no saponification) to 3 (severe saponification)
Change from Baseline in Demodex Presence to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Subjective assessment of the amount of Demodex present at the base of the lashes using slit lamp biomicroscopy and white light illumination.
Change from Baseline in Number of Blocked or Capped Meibomian Glands to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Subjective assessment of the number of blocked or capped Meibomian Glands using slit lamp biomicroscopy and white light illumination.
Change from Baseline in Lid Margin Telangiectasia Grading to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Subjective grading of the amount of telangiectasia at the lid margins using slit lamp biomicroscopy and white light illumination. This grading ranges from 0 with no telangiectasia to 3 with severe telangiectasia.
Change from Baseline in Meibum Expressibility to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Subjective grading of meibum expressibility of lower eyelids using slit lamp biomicroscopy and white light illumination. This grading ranges from 0 with all glands being expressible to 3 with no glands being expressible.
Change from Baseline in Meibum Quality to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Subjective grading of meibum quality of lower eyelids using slit lamp biomicroscopy and white light illumination. This grading ranges from 0 with clear fluid being expressed to 3 with inspissated toothpaste-like expression.
Change from Baseline in Fluorescein Corneal Staining to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Subjective grading of the amount of corneal staining using fluorescein instillation, cobalt blue light illumination and the Oxford grading scale. This ranges from 0 with no staining to 5 with intense staining.
Change from Baseline in Bulbar Conjunctival Staining to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Subjective grading of the amount of bulbar conjunctival staining using fluorescein and lissamine green instillation, white light illumination and the Oxford grading scale. This ranges from 0 with no staining to 5 with intense staining.
Change from Baseline in Lissamine Green Lid Wiper Epitheliopathy to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Subjective grading of the amount of lid wiper epitheliopathy using lissamine green instillation and white light illumination. This grading ranges from 0 with no lid wiper epitheliopathy to 4 with severe lid wiper epitheliopathy.
Change from Baseline in Meibography Meiboscore to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Subjective grading of the amount of Meibomian gland loss using infrared imaging and the Pult meiboscore. This grading ranges from 0 with no gland loss to 4 with severe gland loss (Pult and Reide-Pult, 2013).
Change from Baseline in MMP-9 Tear Concentration to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Measure of matrix metalloproteinase-9 concentration in tears collected with a capillary and measured with a rapid immunoassay test.
Change from Baseline in LTA Tear Concentration to the Final Follow-up 1 Month After Final Treatment Session | Baseline up to 1 month after final treatment session
  Measure of lymphotoxin-A in tears collected with a capillary and measured with a rapid immunoassay test.

CONTACTS AND LOCATIONS:
Overall Officials: James S Wolffsohn, PhD, Study Director — Aston University
Locations (2):
- University of Auckland, Auckland, New Zealand
- Aston Dry Eye Clinic, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Deidentified datasets will be available upon request.
Time Frame: Deidentified datasets will be available upon request.
Access Criteria: Deidentified datasets will be available upon request.

REFERENCES:
- [Background] Tomlinson A, Bron AJ, Korb DR, Amano S, Paugh JR, Pearce EI, Yee R, Yokoi N, Arita R, Dogru M. The international workshop on meibomian gland dysfunction: report of the diagnosis subcommittee. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):2006-49. doi: 10.1167/iovs.10-6997f. Print 2011 Mar. No abstract available. PMID 21450918
- [Background] Pult H, Riede-Pult B. Comparison of subjective grading and objective assessment in meibography. Cont Lens Anterior Eye. 2013 Feb;36(1):22-7. doi: 10.1016/j.clae.2012.10.074. Epub 2012 Oct 27. PMID 23108007
- [Background] Wolffsohn JS, Arita R, Chalmers R, Djalilian A, Dogru M, Dumbleton K, Gupta PK, Karpecki P, Lazreg S, Pult H, Sullivan BD, Tomlinson A, Tong L, Villani E, Yoon KC, Jones L, Craig JP. TFOS DEWS II Diagnostic Methodology report. Ocul Surf. 2017 Jul;15(3):539-574. doi: 10.1016/j.jtos.2017.05.001. Epub 2017 Jul 20. PMID 28736342
- [Background] Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. doi: 10.1001/archopht.118.5.615. PMID 10815152
- [Background] Chalmers RL, Begley CG, Caffery B. Validation of the 5-Item Dry Eye Questionnaire (DEQ-5): Discrimination across self-assessed severity and aqueous tear deficient dry eye diagnoses. Cont Lens Anterior Eye. 2010 Apr;33(2):55-60. doi: 10.1016/j.clae.2009.12.010. Epub 2010 Jan 25. PMID 20093066
- [Background] Arita R, Minoura I, Morishige N, Shirakawa R, Fukuoka S, Asai K, Goto T, Imanaka T, Nakamura M. Development of Definitive and Reliable Grading Scales for Meibomian Gland Dysfunction. Am J Ophthalmol. 2016 Sep;169:125-137. doi: 10.1016/j.ajo.2016.06.025. Epub 2016 Jun 23. PMID 27345733